CLINICAL TRIAL: NCT03869307
Title: Shoulder Exercises in Patients With Hypermobility Spectrum Disorder and Long-lasting Shoulder Symptoms: A Randomised Controlled Trial
Brief Title: Shoulder Exercises in Hypermobile Patients With Shoulder Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Esbjerg Municipality (Other Government); The Danish Rheumatism Association (Other); Region of Southern Denmark (Other); Fund for Research, Quality and Education in Physiotherapy Practice (Unknown)
Responsible Party: Principal Investigator, Behnam Liaghat, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20170066-RCT
Record Dates: First submitted 2019-03-05; First posted 2019-03-11 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Hypermobility Syndrome Shoulder; Shoulder Pain Chronic; Shoulder Luxation
Keywords: Joint instability; Hypermobility; Shoulder; Strength training
MeSH Terms: conditions — Shoulder Dislocation; Joint Instability | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder strengthening exercises (Experimental): Progressive heavy shoulder strengthening exercises three times weekly and advice on load and pain management. Exercise sessions are supervised twice a week corresponding to 32 supervised exercise sessions during the 16 weeks.
  Interventions: Other: Exercise
- Shoulder stability exercises (Active Comparator): Recommendations of shoulder stability exercises which are to be performed unsupervised (e.g. at home) three times weekly and advice on load and pain management. Three supervised sessions are offered during the 16 weeks, and exercises are primarily performed unsupervised at home.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The exercise programme includes exercises identified in literature to target scapular and rotator cuff muscles.

SUMMARY:
Hypermobility Spectrum Disorder (HSD) is a recent diagnosis that covers generalised joint hypermobility with one or more secondary symptomatic musculoskeletal manifestations. Current clinical management of this population with shoulder symptoms is based on limited evidence and includes a combination of non-specific physiotherapy modalities and exercise prescription. There is some evidence suggesting that strength training may be valuable for treatment of this patient-group. Therefore, the aim of this study is to evaluate the effectiveness of a heavy shoulder strengthening exercise programme in patients with HSD and shoulder symptoms.

DETAILED DESCRIPTION:
Hypermobility Spectrum Disorder (HSD) is a recent diagnosis that covers generalised joint hypermobility with one or more secondary symptomatic musculoskeletal manifestations such as chronic shoulder pain and shoulder instability. The evidence for treatment is sparse, but current clinical management of this patient-group with persistent shoulder symptoms is a combination of non-specific physiotherapy modalities and exercise prescription. There is some evidence suggesting that strength training may be valuable for treatment of this patient-group. The intervention consisting of heavy shoulder strengthening exercises has recently been tested to be feasible, and since clinical improvements were seen, the intervention is ready to be studied in a randomised controlled trial. Therefore, the aim of this study is to evaluate the effectiveness of a heavy shoulder strengthening exercise programme and general advice as compared to shoulder stability exercises and general advice (current standard care) in patients with HSD and persistent shoulder symptoms. The primary hypothesis is that a heavy shoulder strengthening exercise programme is superior to standard care.

Sample size considerations: a clinically significant effect of 252 points or more out of 2100 points (SD = 350 points) between the two groups over the 16 weeks is desired, which with a two-sided significance of 0.05, a power of 0.9, and 16% dropout, requires a total of 100 patients. In case 100 patients are not included within 24 months, a stopping rule will be applied as soon as at least 76 patients are included, corresponding to a power of minimum 0.8.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 65
* Generalized HSD (G-HSD) defined with Beighton score cut-off ≥ 5 for women up to the age of 50 years and ≥ 4 for those above 50 years and all men, or Historical HSD (H-HSD) if the Beighton score was 1 point below the age and sex-specific cut-off AND the five-part questionnaire (5PQ) was positive (= at least two positive items).
* Present with one or more secondary symptomatic musculoskeletal manifestations, defined as either

  1. musculoskeletal pain in minimum one shoulder for at least three months

     and/or
  2. recurrent joint dislocations or joint instability without a reported history of trauma defined as either a) minimum three atraumatic dislocations in same shoulder, b) minimum two atraumatic dislocations in two different joints (minimum one in the shoulder) occurring at different times, or c) medical confirmation of joint instability in minimum two joints (minimum one in the shoulder) not related to trauma.

Exclusion Criteria:

* Clinically suspected referred pain from the cervical spine
* Systemic inflammatory rheumatic diseases
* Connective tissue diseases (e.g. Marfans, Stickler's or Loeys Dietz syndromes, Ehlers-Danlos Syndromes except hypermobile type)
* Neurological diseases
* Pregnancy or childbirth within the past year or planning to get pregnant during the study period
* Shoulder surgery within the past year
* Steroid injection in the affected shoulder within three months
* Inability to speak and understand Danish.
* Unable to comply with protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario Shoulder Instability Index (WOSI) questionnaire total score | 16 weeks
  Western Ontario Stability Index questionnaire (WOSI) is a tool designed for self-assessment of shoulder function for patients with instability problems.
  This questionnaire has 21 questions, each scored on a scale from 0 to 100, with 0 being the best score (no limitations related to the shoulder) and 100 representing the worst score. Overall, the questionnaire is scored from 0-2100 points (better to worse).
  There are subscale components reporting on: physical symptoms (questions 1 through 10; maximum score of 1000); sports/recreation/work (questions 11 through 14; maximum score 400); lifestyle (questions 15 through 18; maximum score 400); and emotion (questions 19-21; maximum score 300).
  Subscale scores are added to determine the total score out of a possible 2100 points, with 2100 representing the worst possible score.

SECONDARY OUTCOMES:
Change in pain level on numeric pain rating scale | 12 months.
  Assessment of shoulder pain will be measured by the Numerical Rating scale of pain (NPRS) with numbers from 0 - 10 ("no pain" to "extreme pain"). The pain level will be measured at baseline as the intensity of pain right now, and at 16 weeks follow-up, and in addition, the worst, least and average pain level for the past week will be measured one time weekly.
Change in symptom level on numeric rating scale | 12 months.
  Assessment of shoulder symptoms other than pain (instability, subluxation, looseness) will be measured by the Numerical Rating Scale (NRS) with numbers from 0 - 10 ("no symptoms" to "extreme symptoms"). The symptom level will be measured at baseline as the intensity of symptoms right now, and at 16 weeks follow-up. In addition, the worst, least and average symptoms levels for the latest week will be measured one time weekly.
Change in Checklist Individual Strength (CIS), fatigue subscale | 12 months.
  Assessment of fatigue by the Checklist Individual Strength (CIS), subscale fatigue will be performed at baseline and at 16-week follow up to report the change in level of fatigue. CIS Subscale fatigue consists of 8 items each scored on a 7-point Likert scale (scores ranging from 8 to 56) with high scores indicating high levels of fatigue Timepoints: baseline, 16 weeks, 12 months
Change in Dartmouth Primary Care Cooperative Research Network/World Organization of National Colleges, Academies and Academic Associations of General Practitioners/Family Physicians (COOP/WONCA) | 12 months.
  To assess the change in functional health status from baseline to 16 weeks follow-up the COOP/WONCA questionnaire will be used. The questionnaire is a generic health status questionnaire for General Practice patients. The questionnaire consists of six single-item measures; physical fitness, feelings (mental well-being), daily activities, social activities, besides change in health and overall health. The categories chosen are scored from one (good functional status) to five (poor functional status) (scores ranging from 6-30, best to worse) Timepoints: baseline, 16 weeks, 12 months
Change in Tampa Scale of Kinesiophobia (TSK-11) | 12 months.
  Tampa scale of Kinesiophobia is used to measure impression of change in fear of movement from baseline to 16 weeks follow-up. It consists of an 11-item scale where each question is scored on a 4 point Likert scale, with 1 indicating, "strongly disagree" and 4 indicating, "strongly agree". The total scores range from 11-44, with higher scores representing increased fear of movement.
Change in EuroQol 5 dimension 5 level (EQ-5D-5L) | 12 months.
  The EQ-5D-5L measures change in health related quality of life and includes the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D descriptive system comprises five dimensions (mobility, Self-care, usual activities, pain/discomfort and anxiety/depression). Each dimension is rated using a five-level ordinal scale from no problems to extreme problems. It results in a preference based index that range from states worse than death (<0), to 1 (full health), anchoring dead at 0. A score of one indicates that the participants perceived their health at the best possible state and a score below null that the participants perceived their health worse than death.
  The EQ VAS measures change in health related quality of life. It includes a visual analogue scale where own health 'today´ is rated on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Change in isometric shoulder strength | 16 weeks.
  Maximum isometric voluntary contraction (MVC) in shoulder scaption, internal rotation and external rotation using a hand-held dynamometer (IsoForce Dynometer EVO2; Medical Device Solutions AG).
Change in active and passive shoulder range of motion | 16 weeks
  Internal rotation and external rotation with shoulder in 90 degrees of abduction is measured using a HALO digital goniometer (Halo Medical Devices, Subiaco, Australia).
Change in shoulder proprioception | 16 weeks
  Shoulder proprioception is measured in shoulder flexion angles (low and mid) using af HALO digital goniometer.
Change in Patient Specific Functional Scale (PSFS) | 12 months.
  Patient Specific Functional Scale (PSFS) is administered verbally and used to evaluate whether a health condition impacts a patient's ability to perform activities that are important to him/her. On the initial assessment, the patient is asked to identify up to three important activities that are unable to do or are having difficulty with as a result of symptoms." The patient then provides a rating for each item, on an 11-point ordinal scale ranging from 0 ("unable to perform activity") to 10 ("able to perform activity at the same level as before the injury or problem"). During reassessments, the patient is prompted to re-rate the same activities. The average of up to 3 specific activity scores is recorded, and the range of possible scores is 0 - 10. Higher scores indicate less impairment.
Change in clinical shoulder tests | 16 weeks.
  Joint mobility and laxity parameters are assessed using load and shift, sulcus sign, Gagey, apprehension, relocation, release, Rotés Qúerol shoulder hypermobility test, shoulder flexion hypermobility test, and shoulder rotation hypermobility test, all of which are rated as dichotomous (yes/no).
Adverse events | 12 months.
  Adverse events (AE) and serious adverse events (SAE) will be recorded by a weekly questionnaire and at 16-week and 12-month follow-ups by asking the patients about potential AEs using open-probe questioning to ensure that all AEs are recorded. AEs will be categorized into index shoulder or other sites and will be recorded and assessed for severity independent of whether or not there is a causal relationship with study treatments.
Change in subscales of the Western Ontario Shoulder Instability Index (WOSI) questionnaire | 12 months.
  Western Ontario Stability Index questionnaire (WOSI) is a tool designed for self-assessment of shoulder function for patients with instability problems.
  This questionnaire has 21 questions, each scored on a scale from 0 to 100, with 0 being the best score (no limitations related to the shoulder) and 100 representing the worst score.
  Overall, the questionnaire is scored from 0-2100 points (better to worse). There are subscale components reporting on: physical symptoms (questions 1 through 10; maximum score of 1000); sports/recreation/work (questions 11 through 14; maximum score 400); lifestyle (questions 15 through 18; maximum score 400); and emotion (questions 19-21; maximum score 300).
Physical Activity | Baseline
  The International Physical Activity Questionnaire (IPAQ) is a patient-reported measure of physical activity on a 12-item scale. The total score will be summed within each physical activity domain to estimate the total time spent in occupational, transport, household, and leisure related physical activity, as well as total time reported sitting per week. The total score ranges from 0 to the highest number of time (hours) that the participants can spent on physical activity. A higher score means higher level of physical activity.
Global Perceived Effect (GPE) | 16 weeks
  To measure the patients self-rated impression of improvement at follow-up the GPE will be used related to the WOSI subscales (physical symptoms, sports/recreation/work, lifestyle, and emotions). GPE measures self-rated impression of improvement since baseline assessment on a 7-point scale (1 "worse, an important worsening" to 7 "better, an important improvement)
Compliance with exercise | 16 weeks
  The number of exercise sessions that the patient completes out of 48 sessions.
Demographic | Baseline
  Age, questions regarding civil status, educational level, employment, disease history and previous treatment.
Anthropometrics | Baseline and 16 weeks
  Body mass index

OTHER OUTCOMES:
Patient Acceptable Symptom State (PASS) | 12 months.
  "When you think of your shoulder function, will you consider your current condition as satisfying? By shoulder function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life". Answered by "yes" or "no".
Patient-reported treatment failure | 12 months.
  Only answered by patients answering "no" to PASS. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?". Answered by "yes" or "no".
Change in Pain Self-Efficacy Questionnaire (PSEQ) | baseline
  Patients will be evaluated on self-efficacy related to symptoms, which can be defined as an individual's confidence to successfully produce desirable results related to living with symptoms. The PSEQ has 10 items which are rated on a 7-point ordinal scale (ranging from 0: "not at all confident" to 6: "completely confident"). The maximum score is 60 and higher the score, higher the level of self-confidence of the patient to self-manage their symptoms.
Patient expectations | Baseline
  Patient expectations of treatment effectiveness will be evaluated by asking 'How much do you expect your shoulder problem to change as a result of physiotherapy treatment', measured on a 7-point Likert scale ranging from 0 'worse than ever' to 7 'completely recover'

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Liaghat, MSc, Principal Investigator — University of Sotuhern Denmark; Birgit Juul-Kristensen, PhD, Study Director — University of Southern Denmark; Søren T Skou, PhD, Study Chair — University of Southern Denmark, Næstved-Slagelse-Ringsted Hospitals; Karen Søgaard, PhD, Study Chair — University of Southern Denmark; Jens Søndergaard, MD, PhD, Study Chair — University of Southern Denmark
Locations (3):
- Denmark (3):
  - GPs and physiotherapists, Esbjerg, Region Syddanmark
  - GPs and physiotherapists, Middelfart, Region Syddanmark
  - GPs and physiotherapist, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request after the primary publications have been published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Ultimo 2022
Access Criteria: Data will be made available upon reasonable request after the primary publications have been published.

REFERENCES:
- [Background] Liaghat B, Skou ST, Sondergaard J, Boyle E, Sogaard K, Juul-Kristensen B. A randomised controlled trial of heavy shoulder strengthening exercise in patients with hypermobility spectrum disorder or hypermobile Ehlers-Danlos syndrome and long-lasting shoulder complaints: study protocol for the Shoulder-MOBILEX study. Trials. 2020 Dec 1;21(1):992. doi: 10.1186/s13063-020-04892-0. PMID 33261635
- [Result] Liaghat B, Skou ST, Sondergaard J, Boyle E, Sogaard K, Juul-Kristensen B. Short-term effectiveness of high-load compared with low-load strengthening exercise on self-reported function in patients with hypermobile shoulders: a randomised controlled trial. Br J Sports Med. 2022 Jun 1;56(22):1269-76. doi: 10.1136/bjsports-2021-105223. Online ahead of print. PMID 35649707
- [Result] Liaghat B, Skou ST, Sondergaard J, Boyle E, Sogaard K, Juul-Kristensen B. Clinical Characteristics of 100 Patients With Hypermobility Spectrum Disorders and Shoulder Complaints With or Without Mechanical Symptoms: A Cross-sectional Study. Arch Phys Med Rehabil. 2022 Sep;103(9):1749-1757.e4. doi: 10.1016/j.apmr.2021.12.021. Epub 2022 Jan 21. PMID 35065941
- [Derived] Liaghat B, Juul-Kristensen B, Faber DA, Christensen EO, Sogaard K, Skou ST, Sondergaard J, Juhl CB. One-year effectiveness of high-load compared with low-load strengthening exercise on self-reported function in patients with hypermobile shoulders: a secondary analysis from a randomised controlled trial. Br J Sports Med. 2024 Mar 21;58(7):373-381. doi: 10.1136/bjsports-2023-107563. PMID 38253436
- See also: Protocol paper — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-020-04892-0
- See also: Primary results — https://bjsm.bmj.com/content/early/2022/05/31/bjsports-2021-105223